CLINICAL TRIAL: NCT06538350
Title: Telemedicine in Palliative Care: Interventions, Experiences and Perceptions of Patients Diagnosed With Cancer Receiving Outpatient Palliative Care
Brief Title: Telemedicine in Palliative Care: Interventions, Experiences and Perceptions of Patients Diagnosed With Cancer
Acronym: PALTEL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OncoHelp Association (Other)
Responsible Party: Principal Investigator, Alexandra Kovacs, Principal Investigator, OncoHelp Association
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Telemedicine. Palliative Care.
Record Dates: First submitted 2024-07-25; First posted 2024-08-05 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Advanced Cancer
Keywords: Cancer; Palliative Care; Telemedicine; Outpatient
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, single-centre, randomized, with parallel assignment, controlled trial, with a 1:1 allocation across two treatment arms: telemedicine consultations versus face-to-face consultations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine consultations (Experimental): The experimental intervention will be delivered via Zoom and Video WhatsApp platforms via a secure internet connection.
  Interventions: Other: Telemedicine Consultation
- Face-to-Face Consultations (Active Comparator): Patients randomised to the control arm will continue with face-to-face consultations according to the standard of care.
  Interventions: Other: Face-to-Face Consultation

INTERVENTIONS:
Other: Telemedicine Consultation — Telemedicine intervention will be delivered via Zoom and Video WhatsApp platforms via a secure internet connection.
  Arms: Telemedicine consultations
Other: Face-to-Face Consultation — Face-to-Face consultation according to the standard of care.
  Arms: Face-to-Face Consultations

SUMMARY:
The aim of this study is to estimate the effects of a palliative care consultation intervention among adults with advanced cancer delivered either as a remote (telemedicine) or face-to-face consultation, on changing symptom scores, quality of life, communication, participants' experiences, e-health literacy, emergency and unscheduled visits, adherence to treatment, retention rate, adherence rate, the level of satisfaction of patients and healthcare professionals.

DETAILED DESCRIPTION:
This is a prospective, single-centre, randomized, with parallel assignment, controlled trial, with a 1:1 allocation across two treatment arms: telemedicine consultations versus face-to-face consultations.

All trial activities will be conducted through the Outpatient Clinic of OncoHelp Association located in Timisoara, Romania.

Participants in this study will be recruited from newly diagnosed cancer patients who have not received palliative care interventions prior to enrollment. They are referred to the Outpatient Clinic of the OncoHelp Association for oncological and palliative registration, consultations, and treatment.

After gaining informed consent, a baseline assessment will be collected, including screening feasibility for the telemedicine arm. The selected patients will be randomly allocated with a 1:1 ratio to receive either:

Telemedicine consultation ( Intervention Arm) Group A Face-to-Face consultation ( Control Arm) Group B The participants will receive three monthly consultation and unscheduled consultations as they need according to the study arm they had been allocated.

The participants will benefit from the following categories of interventions depending on their needs :

1. Communication of diagnosis, prognosis, and treatment options
2. Mediation of patient-caregiver communication
3. Symptom control for pain, fatigue, nausea, depression, anxiety, drowsiness, comfort, dyspnoea, sweating, cough, constipation, haemorrhage, itching, secretions, dysphagia, appetite
4. Care of wounds, bedsores, stomas
5. End of life care
6. Patient and caregiver education
7. Psychological counseling
8. Reports for obtaining social rights (sickness pension, disability pension)
9. Reports for obtaining devices provided without personal contribution by the health insurance system
10. Referral for spiritual assistance
11. Management plan
12. Referral for specialized service level III
13. Referral for hospitalization
14. Unscheduled consultations

ELIGIBILITY:
Inclusion Criteria:

Participant Inclusion Criteria

* Adult patients, age ≥ 18 years
* Diagnosis of solid tumour in any stage, regardless of location
* Participant diagnosed within the last 90 days with advanced or metastatic cancer (defined as a newly diagnosed stage II-IV, recurrence, or progressive solid tumour cancer)
* Eastern Cooperative Oncology Group (ECOG ) 1 ( ambulatory ) - 3 ( symptomatic, bed immobilised> 50% during the day )
* Estimated life expectancy of at least three months
* Participants can receive any cancer treatment for their advanced cancer while participating in this study
* Receiving primary cancer care at the participating site
* Have access to a telephone that can receive incoming calls
* Participant/ caregiver can use a personal computer, smartphone, tablet
* Participants must have access to a Wi-Fi network or a cellular network
* Participant can communicate verbally
* Participant can read and respond to questions in the Romanian language
* Participant able to provide informed consent
* Participant has a considerable disease burden and complex medical and care needs
* Participant is at a medium to high risk of worsening their condition, requiring hospitalisation, or having an increased need for health and care services
* Participant has a high consumption of healthcare services
* Participant has a reduced level of function
* Participant is motivated to use telemedicine and will likely benefit from telemedicine solutions
* Participant are willing to adhere to telemedicine consultations or face-to-face consultations

Caregiver Inclusion Criteria

* Adult , age ≥ 18 years
* Relative or friend who is identified by the Participant and lives with the Participant or has contact with him/her at least twice per week
* The ability to read and respond to questions in Romanian language
* Caregiver who is willing to participate in the study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Have not themselves been diagnosed with cancer or received cancer treatment during the study (to ensure that the Participant and the caregiver focus their efforts on the care of the Participant)
* Caregiver must have access to a computer/ tablet/ smartphone and an internet connection at home, on which they would be willing to do a telemedicine study
* Be able to navigate websites, communicate by email, and have regular access to the internet (assessed by participant self-report)
* Be capable of independently utilising an online platform for telemedicine medical consultations in a private setting (assessed by participant self-report)

Exclusion Criteria:

Participant Exclusion Criteria

* Participant already receiving outpatient palliative care or hospice services
* Participant with Eastern Cooperative Oncology Group (ECOG) 4 performance status
* Participant too medically unstable (or expected to become so during the study period) to participate in a telemedicine group medical visit determined by the investigator
* Participants with a high level of distress who cannot be managed by telemedicine
* End of Life
* Participant with extensive hearing loss such that the ability to participate in the study would be impaired as determined by the investigator
* Self-reported history of a diagnosis of dementia
* Self-reported psychotic symptoms in the last 30 days prior to randomisation
* Active suicidal ideation (currently reported suicidal plan and intent)
* Self-reported active alcohol or substance abuse in the last 30 days prior to randomisation
* Any change in psychotropic medications within the last 30 days
* Participant without medical insurance that covers telemedicine consultations or face-to-face consultations
* Participant who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* Failure/inability/unwillingness to provide names and contact information for two family members or friends to serve as emergency contacts during the study

Caregiver Exclusion Criteria

* Adult caregiver, age ≥ 18 years
* Cognitive or psychiatric conditions as determined by the researcher investigator to prohibit study participation
* Non-compliant caregiver with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Patients' Quality of Life . | 12 weeks
  To determine whether telemedicine palliative care consultations are equivalent to face-to-face palliative care consultations for improving patients' quality of life as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire(EORTC-QLQ-C30). All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
  Patients' Quality of Life [ Time Frame:12 weeks] To determine whether telemedicine consultations palliative care is are equivalent to face-to-face palliative care consultations for improving patients' quality of life as measured by the EORTC-QLQ-C30 Questionnaire.
Changes in symptom control . | 12 weeks
  Symptom management will be measured through the mean changes in distress score on the Integrated Palliative care Outcome Scale (IPOS). There are 10 questions scored on a scale of 1-4, which assess a patient's symptoms and needs with regards to physical, social, psychological and spiritual. Individual IPOS item scores of zero or one require less clinical attention than items that score three or four.
Patients' satisfaction . | 12 weeks
  To assess the effect of the superiority of telemedicine versus face-to-face consultations about palliative care on patient satisfaction as measured by the 16-item measure of Patient Satisfaction Questionnaire(FAMCARE P 16 Questionnaire). This is a self-report scale assessing patient satisfaction with outpatient palliative oncology care, which is composed of 16 items rated from 1 (very dissatisfied) to 5 (very satisfied). Higher scores are related to higher satisfaction with the care received.

SECONDARY OUTCOMES:
eHealth Literacy . | Baseline and 12 weeks after baseline
  Participants' ability to find and evaluate online health information will be measured using the eHealth Literacy Scale. The eHealth literacy scale is an eight-item scale used to asses self-reported capability of eHealth consumers to find, appraise, and use health related information from the internet to solve health problems . Scores are interpreted as follows: Predominantly Disagree: Scores range from 8 to 15.99; Mostly Disagree: Scores range from 16 to 23.99. Mostly Agree: Scores range from 24 to 31.99. Predominantly Agree: Scores range from 32 to 40.
Domain of intervention . | 12 weeks
  The interventions provided in this study will respect the principle of holistic care. Depending on the patient's needs, interventions will be provided in the physical, emotional, social, and spiritual domains during each scheduled or unscheduled visit.
  During each visit, the interventions granted and the domains - physical, emotional, social and spiritual - to which these interventions belong will be recorded.
Number of patients satisfied with physician communication . | 12 weeks
  14-item Communication Assessment Tool (CAT) will be used. The CAT specifically addresses patient satisfaction with key aspects of communication and interpersonal skills, and items are scored on a 1-5 scale where 1 = poor and 5 = excellent, and a higher score would indicate better communication skills.
Patients' experiences . | 12 weeks
  Participants' experiences with the care will be measured using the Patient Reported Experience Measures Questionnaire (PREMs). Patients' experience is rated from poor (rated as 1) to excellent (rated as 5). Higher scores are related to higher satisfaction during consultation.
Number of emergency room visit . | 12 weeks
  Monitoring patient interactions with the Emergency Room (ER) during the trial period.
Number of unscheduled visits . | 12 weeks
  Monitoring the number of unscheduled visits.
Adherence to intervention . | 12 weeks
  Intervention adherence will be estimated as the mean proportion of the scheduled consultations each participant completes .
Changes in medication adherence . | 12 weeks
  Medication adherence will be measured using the Morisky Medication - Taking Adherence Scale (MMAS-4 Scale). The MMAS consists of four items, with a scoring scheme of "Yes" = 0 and "No" = 1. The items are summed to give a range of scores from 0 to 4 .
Number of completed telemedicine scheduled visits . | 12 weeks
  Telemedicine will be feasible in this population if at least 80% complete the telemedicine visits. A visit will be considered successful if all measurements are recorded.
Physicians ability to evaluate a patient through telemedicine . | 12 weeks
  Measured by the Provider Satisfaction with Telemedicine Questionnaire. This questionnaire will be completed by the interventionists after visit 3 . This survey included included 5 components: demographics, care settings, experience, motivation, and overall satisfaction.

OTHER OUTCOMES:
Proportion of participants enrolled | Baseline
  The proportion of eligible and approached patients who consent to participate.
Number of participants ineligible or refusing to participate . | Baseline
  Number of participants who are determined to be ineligible before the first visit.
Frequency of participant ineligibility reason | Baseline
  Potential study candidates who are ineligible will be recorded for reasons of ineligibility.
Frequency of participant refusal reason | Baseline
  Potential study candidates who decide not to participate will be recorded for refusal reasons.
Retention rate | 12 weeks
  The percentage of patients who remained in the study and did not drop out of their own accord.
Completion rate | 12 weeks
  The percentage of patients who completed the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kovacs, MD, Study Chair — OncoHelp Association

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kovacs A, Payne S, Mosoiu D. Efficacy of telemedicine for cancer patients in outpatient palliative care setting: Protocol of a randomized, open-label, non-inferiority study. Palliat Care Soc Pract. 2026 Jan 13;20:26323524251408888. doi: 10.1177/26323524251408888. eCollection 2026. PMID 41550463